CLINICAL TRIAL: NCT06436781
Title: Effect of Maolactin™ FMR Supplementation on Exercise Recovery, Inflammation, and Muscle Comfort in an Otherwise Healthy Population: A Double-blind Randomized Placebo-controlled Study
Brief Title: Effect of Maolactin™ FMR on Exercise Recovery, Inflammation, and Muscle Comfort in an Otherwise Healthy Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAOJOI(A)
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-10

CONDITIONS: Post Exercise Inflammation; Exercise Recovery; Muscle Fatigue; Muscle Pain
MeSH Terms: conditions — Myalgia | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maolactin (Experimental): 2 capsules containing a total of 500 mg/day active proteins taken once daily before the morning meal
  Interventions: Drug: Maolactin
- Maltodextrin (Placebo Comparator): 2 capsules containing maltodextrin (0mg/day active proteins) taken once daily before the morning meal
  Interventions: Drug: Maltodextrin

INTERVENTIONS:
Drug: Maolactin — Once daily dose of 2 capsules containing a total of 500mg/day Maolactin
  Arms: Maolactin
Drug: Maltodextrin — Once daily dose of 2 capsules of Maltodextrin containing a total of 0mg/day Maolactin
  Arms: Maltodextrin

SUMMARY:
This is a double blind, randomised, placebo-controlled, parallel-group trial to evaluate the effect of Maolactin FMR supplementation on post exercise inflammation, exercise recovery and muscle fatigue and pain in an otherwise healthy population of adults 18-65 years old over 10 weeks with 8 weeks of supplementation.

This is PART A of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years old
* Generally healthy
* BMI 19.0 - 29.9 kg/m2
* Able to provide informed consent
* Generally active, low to moderately trained (with a minimum of 1 resistance exercise sessions per week)
* Agree not to change current diet and/or exercise frequency or intensity during study period
* Agree to not participate in another clinical trial while enrolled in this trial

Exclusion Criteria:

* Undertaking high intensity exercise training and or undertaking more than 3 days of resistance training per week.
* Serious illness(1) e.g., mood disorders such as depression, anxiety or bipolar disorder, neurological disorders such as MS, kidney disease, liver disease or heart conditions
* Unstable illness(2) e.g., diabetes and thyroid gland dysfunction
* Unstable intake of any medication or supplement(3)
* Acute injuries on reporting area
* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy including low dose aspirin
* Receiving medications known to affect inflammation such as steroids
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>21 alcoholic drinks per week)
* Pregnant or lactating women
* Allergic to any of the ingredients in active or placebo formula
* Participants who are currently participating in any other clinical trial or who have participated in any other clinical trial during the past 1 month
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion

  1. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.
  2. An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity.
  3. An unstable intake is any dose that has changed by more than 10% of the previous dose in the past 4-weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Change in post exercise muscle breakdown | Baseline (Pre-exercise and 0, 1, 2, 24 and 48 hours post exercise) and Week 8 (Pre-exercise and 0, 1, 2, 24 and 48 hours post exercise)
  Change in post exercise muscle breakdown as assessed by creatine kinase (CK) via blood test

SECONDARY OUTCOMES:
Change in Weight | Baseline and Week 8
  Change in Weight as measured by digital scales
Change in Body Mass Index (BMI) | Baseline and Week 8
  Change in BMI as assessed by digital scale for weight and stadiometer for height
Change in Musculoskeletal Health Questionnaire (MSK-HQ) | Baseline (Session 1, Session 2 (+24 hours), Session 3 (+48 hours)) and Week 8 (Session 1, Session 2 (+24 hours), Session 3 (+48 hours))
  Change in MSK-HQ as self-reported by participants. Scored on a range of 0-56, with a higher score indicating health status.
Change in Visual Analogue Scale (VAS) Muscle Pain | Baseline (Session 1, Session 2 (+24 hours), Session 3 (+48 hours)) and Week 8 (Session 1, Session 2 (+24 hours), Session 3 (+48 hours))
  Change in VAS Muscle Pain as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of muscle pain.
Change in Visual Analogue Scale (VAS) Pain | Baseline (Session 1, Session 2 (+24 hours), Session 3 (+48 hours)) and Week 8 (Session 1, Session 2 (+24 hours), Session 3 (+48 hours))
  Change in VAS Pain as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of pain
Change in Visual Analogue Scale (VAS) Fatigue | Baseline (Session 1, Session 2 (+24 hours), Session 3 (+48 hours)) and Week 8 (Session 1, Session 2 (+24 hours), Session 3 (+48 hours))
  Change in VAS Fatigue as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of fatigue.
Change in Visual Analogue Scale (VAS) Mobility | Baseline (Session 1, Session 2 (+24 hours), Session 3 (+48 hours)) and Week 8 (Session 1, Session 2 (+24 hours), Session 3 (+48 hours))
  Change in VAS Mobility as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of mobility.
Change in Visual Analogue Scale (VAS) Stiffness | Baseline (Session 1, Session 2 (+24 hours), Session 3 (+48 hours)) and Week 8 (Session 1, Session 2 (+24 hours), Session 3 (+48 hours))
  Change in VAS Stiffness as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of stiffness.
Change in Multidimensional Fatigue Inventory (MFI) | Baseline (Session 1, Session 2 (+24 hours), Session 3 (+48 hours)) and Week 8 (Session 1, Session 2 (+24 hours), Session 3 (+48 hours))
  Change in MFI as self-reported by participants. Comprises 20 questions rated on a 5 point scale. with a higher score indicating a higher level of fatigue.
Change in The Perceived Recovery Status Scale (PRSS) | Baseline (Session 1, Session 2 (+24 hours), Session 3 (+48 hours)) and Week 8 (Session 1, Session 2 (+24 hours), Session 3 (+48 hours))
  Change in PRSS as self-reported by participants. A single-item, 0 to 10 point scale where 0 = very poorly recovered (poor performance) and 10 = fully recovered (optimal performance).
Change in Blood Pressure (BP) | Baseline and Week 8
  Change in BP as assessed by digital blood pressure monitor
Change in Heart Rate (HR) | Baseline (Time 0 and every 5 minutes until return to baseline) and Week 8 (Time 0 and every 5 minutes until return to baseline)
  Change in HR as assessed by digital heart rate monitor
Change in Oxygen Saturation | Baseline and Week 8
  Change in Oxygen Saturation as measured by pulse oximeter
Change in Cytokines | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in Cytokines as measured by blood test
Change in Nuclear Factor KappaB (NF-kB) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in NF-kB as measured by blood test
Change in P-selectin | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in P-selectin as measured by blood test
Change in E-selectin | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in E-selectin as measured by blood test
Change in Lipoprotein-associated Phospholipase A2 (Lp-PLA2) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in Lp-PLA2 as measured by blood test
Change in Intercellular Cell Adhesion Molecule-1 (ICAM-1) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in ICAM-1 as measured by blood test
Change in Intercellular Cell Adhesion Molecule-2 (ICAM-2) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in ICAM-2 as measured by blood test
Change in Vascular Cell Adhesion Molecule-1 (VCAM-1) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in VCAM-1 as measured by blood test
Change in Platelet Endothelial Cell Adhesion Molecule-1 (PECAM-1) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in PECAM-1 as measured by blood test
Change in Erythrocyte Sedimentation Rate (ESR) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in ESR as measured by blood test
Change in Lactate Dehydrogenase (LDH) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in LDH as measured by blood test
Change in P38 Mitogen-activated Protein Kinases (P38) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in P38 as measured by blood test
Change in Electrolytes and Liver Function Tests (E/LFT) | Baseline (Pre-exercise and 2 hours post) and Week 8 (Pre-exercise and 2 hours post)
  Change in E/LFT as measured by blood test
Change in Lactic acid | Baseline (Pre-exercise and 0, 1, 2, 24 and 48 hours post exercise) and Week 8 (Pre-exercise and 0, 1, 2, 24 and 48 hours post exercise)
  Change in Lactic acid as measured by blood test
Change in C-reactive protein (CRP) | Baseline (Pre-exercise and 0, 1, 2, 24 and 48 hours post exercise) and Week 8 (Pre-exercise and 0, 1, 2, 24 and 48 hours post exercise)
  Change in CRP as measured by blood test
Change in myoglobin | Baseline (Pre-exercise and 0, 1, 2, 24 and 48 hours post exercise) and Week 8 (Pre-exercise and 0, 1, 2, 24 and 48 hours post exercise)
  Change in myoglobin as measured by blood test
Change in 1 Repetition Max (1-RM) | Baseline (Session 1 and Session 2 (+24 hours)) and Week 8 (Session 1, Session 2 (+24 hours))
  Change in 1 Repetition Max (1-RM) as assessed by exercise testing
Change in Number of Repetitions to Fatigue | Baseline (Session 1 and Session 2 (+24 hours)) and Week 8 (Session 1, Session 2 (+24 hours)
  Change in Number of Repetitions to Fatigue as assessed by exercise testing
Change in Hand Grip Strength | Baseline (Session 1, Session 2 (+24 hours), Session 3 (+48 hours)) and Week 8 (Session 1, Session 2 (+24 hours), Session 3 (+48 hours))
  Change in Hand Grip Strength as measured by dynamometer
Change in BORG Perception of intensity (RPE) | Baseline (Session 1 and Session 2 (+24 hours)) and Week 8 (Session 1, Session 2 (+24 hours)
  Change in BORG Perception of intensity (RPE) as self-reported by participants. Rates exertion from a scale of 6 (no exertion) to 20 (maximum effort). A rating between 12 to 14 typically reflects a moderate or somewhat hard level of intensity.
Change in Adverse Events | 8 week period from enrolment to participant conclusion
  Change in Adverse Events self-reported by participants
Change in Gastrointestinal Tolerance | 1 week after starting product
  Change in Gastrointestinal Tolerance as measured by Gastrointestinal Tolerance (GIT) Questionnaire
Change in diet | Baseline and Week 8
  Change in diet as assessed by 3 day Diet Recall

CONTACTS AND LOCATIONS:
Overall Officials: David Briskey, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Clinical Pty Ltd, Brisbane, Queensland, Australia